CLINICAL TRIAL: NCT05297682
Title: Effects of Repeated Propofol Intravenous Anesthesia on the Postoperative Neurological Function of Patients Undergoing Hysteroscopic Surgery: A Prospective Cohort Study
Brief Title: Effects of Repeated Intravenous Anesthesia With Propofol on the Postoperative Neurological Function of Patients Undergoing Hysteroscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: Liaoqinzff
Record Dates: First submitted 2022-02-28; First posted 2022-03-28 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-02

CONDITIONS: PND; Anesthesia
Keywords: PND
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- singal group: Patients receiving less than two anesthesia in a year
  Interventions: Device: anesthesia with propofol
- repeat group: Patients who received two or more anesthesia in a year
  Interventions: Device: anesthesia with propofol

INTERVENTIONS:
Device: anesthesia with propofol — General anesthesia with propofol

SUMMARY:
Perioperative neurocognitive disorders（PND） is a common complication during the perioperative period, which affects the patient's rehabilitation and quality of life. Animal studies have found that repeated anesthesia and operation lead to neurological disorders. However, there is currently a lack of clinical studies on the effects of repeated anesthesia on patients' neurological function. With the full liberalization of China's three-child policy, the number of women in need of childbearing has increased, and infertile women who repeatedly undergo hysteroscopic surgery under intravenous anesthesia is increasing . Therefore, it is of great significance to investigate whether repeated and repeated general anesthesia and hysteroscopic surgery affect the patient's neurological function. The purpose of this study is to explore the effect of repeated propofol intravenous anesthesia on the neurological function of patients undergoing hysteroscopic surgery.

DETAILED DESCRIPTION:
Central nervous system dysfunction is a common complication during the perioperative period, which affects the patient's rehabilitation and quality of life. Animal studies have found that repeated and multiple anesthesia operations can lead to neurological disorders. However, there is currently a lack of relevant clinical studies on the effects of multiple anesthesia operations on the neurological function of patients. With the full liberalization of China's family planning policy, the number of women in need of childbearing has increased, and the number of patients who repeatedly undergo hysteroscopic surgery under intravenous anesthesia due to infertility in the short term is increasing day by day. Therefore, it is of great significance to investigate whether repeated and repeated general anesthesia and hysteroscopic surgery affect the function of the patient's central nervous system.

Propofol and central nervous system dysfunction during perioperative period Perioperative neurocognitive disorders (PND) include neurocognitive disorders, sleep disorders, and anxiety and depression. The incidence rate is as high as 15%-78%, which affects the rehabilitation and quality of life of patients. A large number of studies have shown that a single anesthesia operation has a slight and short-term impact on the patient's neurological function. However, the impact of multiple anesthesia operations on the patient's neurological function is currently unclear.

Propofol was marketed in the UK in 1986, and was approved in the United States in 1989. It was approved for clinical use in my country in 1994, becoming a widely used clinical general anesthesia induction and maintenance drug. Animal experiments have found that a single exposure of propofol can cause transient neuronal apoptosis and defects in rats, while multiple exposures of propofol can lead to sustained neuronal apoptosis, neuronal defects, synaptic loss, and long-term Cognitive impairment. Repeated exposure to propofol in the neonatal period of rats can damage hippocampal synaptic plasticity and decline in cognitive function in adulthood. Repeated use of propofol can activate the NF-κB pathway and NLRP3 inflammasome, up-regulate the RAGE protein and other pathways, causing hippocampal inflammation and neuronal apoptosis, thereby impairing the cognitive function of elderly rats. The results of these animal studies suggest that repeated and multiple anesthesia operations can lead to neurological disorders. Clinical studies have reported that after a single propofol anesthesia in elderly patients undergoing laparoscopic surgery, 16.8%-18% of patients developed postoperative cognitive dysfunction 7 days after surgery; but whether repeated propofol anesthesia affects the patient's There is no research report on nerve function.

Intrauterine adhesions and transcervical resection of adhesion The infertility rate in China is currently as high as 12.5%-15%, and the number of patients exceeds 50 million, that is, 1 in every 8 couples has infertility problems. intrauterine adhesions (IUA) is a common gynecological uterine disease that seriously harms fertility and has poor treatment effects. It has become the main cause of secondary infertility in Chinese women. Transcervical resection of adhesion (TCRA) is the first choice for infertile women with fertility requirements to treat IUA. However, a large number of literature reports that the re-adhesion rate after TCRA is 30% in mild to moderate IUA, and as high as 62.5% in severe IUA, and the pregnancy success rate is only 22.5%-33.3%. Therefore, due to infertility, many women undergo repeated hysteroscopic surgery under general anesthesia in a short period of time, and some patients have undergone more than 10 anesthesia operations in just 2 years.

With the liberalization of China's plans to formulate policies, the number of patients with secondary infertility who have clinical needs continues to increase. Doctors have always paid more attention to the effect of increasing the uterine cavity of infertile patients, and the story of the neuronal function that may exist in such patients. Therefore, the change describes the clinical treatment plan for the actual infertility patients who have received general anesthesia and hysteroscopic surgery for many times. It is of great significance to social and economic development.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of intrauterine adhesions
* Need hysteroscopic surgery due to intrauterine adhesions
* Women of childbearing age who wish to have children

Exclusion Criteria:

* Those with contraindications to general anesthesia or those who had a history of anesthesia accident
* Those who are known or suspected to be allergic or contraindicated to propofol injection excipients
* Patients with acute upper respiratory tract infection, asthma attack, or acute severe laryngeal disease
* History of gastrointestinal disease: gastrointestinal retention, active bleeding, which may lead to reflux aspiration, etc.
* Complicated medical history of craniocerebral injury, intracranial hypertension, stroke, cerebrovascular accident
* Respiratory insufficiency, obstructive pulmonary disease
* Uncontrolled hypertension, hypotension, and diabetes
* Severe arrhythmia, heart failure, unstable angina, myocardial infarction
* Severe liver dysfunction or severe renal insufficiency
* History of alcoholism or drug dependence
* Abuse or long-term use of narcotic, sedative, and analgesic drugs
* Those who have a history of mental illness
* Participated in any other clinical investigators within 1 month before screening
* Subjects who are considered by the investigator to have any other factors that are not suitable for participating in this research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The enrolled patients who were willing to give birth to undergo hysteroscopic surgery under intravenous general anesthesia were treated with the same protocol of propofol intravenous anesthesia, and the effects of different anesthesia times on the clinical endpoint were compared.
Sampling Method: Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 2 months
  Measured by Montreal cognitive assessment(MoCA)score.The maximum score is 30 points. Lower scores mean worse cognitive function.

SECONDARY OUTCOMES:
Sleep assessment | 1day, 2months
  Measured by The Pittsburgh Sleep Quality Index（PSQI ）score.The PSQI global score has a range of 0-21 points.
Post-operative pain level | 1day, 2 months
  Measured by A numerical rating scale(NRS) score. Score range form 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Postoperative nausea and/or vomiting (PONV) | 1day
  Measured by postoperative nausea and/or vomiting (PONV) yes/no (either by chart or by patient confirmation)
Anxiety level | 1day, 2 months
  Measured by Generalized Anxiety Disorder, (GAD7), GAD-7 total score for the seven items ranges from 0 to 21.0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Depression level | 1day, 2 months
  Measured by Patient Health Questionnaire-9 (PHQ-9).Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Liao, M.D, Principal Investigator — The Third Xiangya Hospital, Central South University
Locations (1):
- The Third Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belrose JC, Noppens RR. Anesthesiology and cognitive impairment: a narrative review of current clinical literature. BMC Anesthesiol. 2019 Dec 27;19(1):241. doi: 10.1186/s12871-019-0903-7. PMID 31881996
- [Background] Lee WL, Liu CH, Cheng M, Chang WH, Liu WM, Wang PH. Focus on the Primary Prevention of Intrauterine Adhesions: Current Concept and Vision. Int J Mol Sci. 2021 May 13;22(10):5175. doi: 10.3390/ijms22105175. PMID 34068335
- [Background] Tasbihgou SR, Absalom AR. Postoperative neurocognitive disorders. Korean J Anesthesiol. 2021 Feb;74(1):15-22. doi: 10.4097/kja.20294. Epub 2020 Jul 6. PMID 32623846
- [Background] Teng Y, Ou M, Wang X, Zhang W, Liu X, Liang Y, Li K, Wang Y, Ouyang W, Weng H, Li J, Yao S, Meng J, Shangguan W, Zuo Y, Zhu T, Liu B, Liu J. Efficacy and safety of ciprofol for the sedation/anesthesia in patients undergoing colonoscopy: Phase IIa and IIb multi-center clinical trials. Eur J Pharm Sci. 2021 Sep 1;164:105904. doi: 10.1016/j.ejps.2021.105904. Epub 2021 Jun 8. PMID 34116176
- [Background] Zhou Z, Zheng D, Wu H, Li R, Xu S, Kang Y, Cao Y, Chen X, Zhu Y, Xu S, Chen ZJ, Mol BW, Qiao J. Epidemiology of infertility in China: a population-based study. BJOG. 2018 Mar;125(4):432-441. doi: 10.1111/1471-0528.14966. Epub 2017 Dec 28. PMID 29030908